CLINICAL TRIAL: NCT04177810
Title: A Phase 2 Study of Plerixafor and Cemiplimab in Metastatic Pancreatic Cancer
Brief Title: Plerixafor and Cemiplimab in Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Genzyme, a Sanofi Company (Industry); American Association for Cancer Research (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J19113; IRB00225153 (Other: Johns Hopkins Medicine Institutional Review Board); 5P01CA247886 (NIH)
Record Dates: First submitted 2019-11-22; First posted 2019-11-26 (Actual); Results first posted 2024-02-20 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Metastatic Pancreatic Cancer
Keywords: Plerixafor; Cemiplimab; Immunotherapy; PD-L1 (receptor blocking antibody); Anti-PD-L1; CXCR4 (chemokine receptor); Antibodies; Metastatic pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — cemiplimab; plerixafor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cemiplimab and Plerixafor (Experimental): All participants will receive Cemiplimab and Plerixafor.
  Interventions: Drug: Cemiplimab; Drug: Plerixafor

INTERVENTIONS:
Drug: Cemiplimab — Cemiplimab (350 mg) will be administered IV on day 1 of each cycle (21 day cycle) for up to 2 years.
  Other Names: REGN-2810, LIBTAYO
Drug: Plerixafor — Plerixafor (80mcg/kg/hr) will be administered as a continuous IV infusion of the first 7 days of each cycle (21 day cycle) for up to 2 years.
  Other Names: AMD3100, MOZOBIL

SUMMARY:
The purpose of this study is to evaluate the safety and clinical activity of plerixafor in combination with cemiplimab in patients with metastatic pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

Age ≥18 years.

* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Have histologically or cytologically-proven ductal pancreatic cancer.
* Have metastatic disease.
* Have documented radiographic disease progression after previous systemic chemotherapy given in a neoadjuvant, adjuvant, locally advanced or metastatic setting.
* Patients with the presence of at least one measurable lesion.
* Willing to have to a tumor biopsy.
* Life expectancy of greater than 3 months.
* Patients must have adequate organ and marrow function defined by study - specified laboratory tests.
* Woman of childbearing potential must have a negative pregnancy test and follow contraceptive guidelines as defined per protocol.
* Men must use acceptable form of birth control while on study.
* Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

* Known history or evidence of brain metastases.
* Had chemotherapy, radiation, or steroids within 14 days prior to study treatment.
* Have received any investigational drugs, a live vaccine, any allergen hyposensitization therapy, growth factors or major surgery within 28 days prior to study treatment.
* Require any antineoplastic therapy.
* Had surgery within 28 days of dosing of investigational agent.
* Has received any prophylactic vaccine within 14 days of first dose of study drug.
* History of prior treatment with anti-CXCR4.
* Have used any systemic steroids within 14 days of study treatment.
* Patients receiving growth factors including, but not limited to, granulocyte-colony stimulating factor (G-CSF), Granulocyte-macrophage colony-stimulating factor (GM-CSF), erythropoietin, within 14 days of study drug administration.
* Hypersensitivity reaction to any monoclonal antibody.
* Evidence of clinical or radiographic ascites.
* Have clinically significant and/or malignant pleural effusion.
* Patient with uncontrolled intercurrent illness including, but not limited to, uncontrolled infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Has an active known or suspected autoimmune disease.
* Prior tissue or organ allograft or allogeneic bone marrow transplantation.
* All toxicities attributed to prior anti-cancer therapy other than alopecia and fatigue must have resolved to grade 1 (National Cancer Institute Common Terminology Criteria for Adverse Events [CTCAE], version 5) or baseline before administration of study drug.
* Infection with HIV or hepatitis B or C at screening.
* Patient has a pulse oximetry of <92% on room air.
* Patient is on supplemental home oxygen.
* Has uncontrolled intercurrent acute or chronic medical illness or any use of illicit drugs or substance abuse.
* Patient is unwilling or unable to follow the study schedule for any reason.
* Woman who are pregnant or breastfeeding.
* Have rapidly progressing disease, as judged by the investigator.
* History of significant, recurrent, unexplained postural hypotension in the last 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2023-03-29 (Actual); Study Completion 2023-05-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dung Le, MD, Principal Investigator — Johns Hopkins Medical Institution
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 4 participants were excluded from analysis because they did not receive at least one dose of study drug.
Groups:
- Cemiplimab and Plerixafor: All participants will receive Cemiplimab and Plerixafor.
  Cemiplimab (350 mg) will be administered IV on day 1 of each cycle (21 day cycle) for up to 2 years.
  Plerixafor (80mcg/kg/hr) will be administered as a continuous IV infusion of the first 7 days of each cycle (21 day cycle) for up to 2 years.
Period: Overall Study
Arm/Group | Cemiplimab and Plerixafor
Started (Started = enrolled and received at least one dose of study drug) | 21
Completed | 20
Not Completed | 1

BASELINE CHARACTERISTICS:
Population: 4 participants were excluded from analysis because they did not receive at least one dose of study drug.
Arm/Group | Cemiplimab and Plerixafor
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) Using Immune RECIST (iRECIST) Criteria
Description: ORR is defined as the number of patients achieving a complete response (CR) or partial response (PR) based on immune Response Evaluation Criteria in Solid Tumors (iRECIST) at any time during the study. CR = disappearance of all target lesions, PR is =>30% decrease in sum of diameters of target lesions, progressive disease (PD) is >20% increase in sum of diameters of target lesions, stable disease (SD) is <30% decrease or <20% increase in sum of diameters of target lesions.
Time Frame: 10 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cemiplimab and Plerixafor
Number analyzed (Participants) | 21
Participants | 0

2. Secondary Outcome: Overall Response Rate (ORR) Using RECIST 1.1 Criteria
Description: Objective Response Rate (ORR) is defined as the number of patients achieving a complete response (CR) or partial response (PR) based on RECIST 1.1 criteria. CR = disappearance of all target lesions, PR is =>30% decrease in sum of diameters of target lesions. Subjects who discontinue due to toxicity or clinical progression prior to post-baseline tumor assessments will be considered as non-responders.
Time Frame: 10 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cemiplimab and Plerixafor
Number analyzed (Participants) | 21
Participants | 0

3. Secondary Outcome: Number of Participants Experiencing Grade 3 or Above Drug-related Toxicities
Description: Defined using NCI CTCAE v5.0
Time Frame: 13 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cemiplimab and Plerixafor
Number analyzed (Participants) | 21
Participants | 4

ADVERSE EVENTS:
Time Frame: Up to 17 months
Description: Serious and Other (Not Including Serious) Adverse Events were evaluated for up to 13 months. All-cause mortality was evaluated for up to 17 months.
Arm/Group | Cemiplimab and Plerixafor
All-Cause Mortality (participants affected / at risk) | 21/21
Serious Adverse Events (participants affected / at risk) | 13/21
Other Adverse Events (participants affected / at risk) | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cemiplimab and Plerixafor (N=21)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Bile Duct Stenosis (Hepatobiliary disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Delerium (Psychiatric disorders) | 1 (1)
Disease Progression (General disorders) | 8 (8)
Fever (General disorders) | 3 (3)
Immune-Mediated Hepatitis (Hepatobiliary disorders) | 1 (1)
Lactic Acidosis (General disorders) | 1 (1)
Lower Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Stroke (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cemiplimab and Plerixafor (N=21)
Abdominal Distension (Gastrointestinal disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 5 (6)
Alanine Aminotransferase Increased (Investigations) | 4 (5)
Alkaline Phosphatase Increased (Investigations) | 6 (7)
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 9 (33)
Anorexia (Metabolism and nutrition disorders) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Ascites (Gastrointestinal disorders) | 1 (1)
Aspartate Aminotransferase Increased (Investigations) | 4 (5)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Bacteremia (Infections and infestations) | 1 (1)
Blood Bicarbonate Decreased (Investigations) | 1 (1)
Blood Bilirubin Increased (Investigations) | 3 (5)
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 3 (3)
Cardiac Troponin I Increased (Investigations) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 8 (11)
Dizziness (Nervous system disorders) | 6 (6)
Dry Mouth (Gastrointestinal disorders) | 2 (2)
Dysesthesia (Nervous system disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 2 (2)
Ear and Labyrinth Disorders (Altered Balance) (Ear and labyrinth disorders) | 1 (1)
Edema Limbs (General disorders) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Fatigue (General disorders) | 3 (4)
Fever (General disorders) | 7 (13)
Flatulence (Gastrointestinal disorders) | 1 (1)
Gastrointestinal Disorders- Melena (Gastrointestinal disorders) | 2 (2)
Hallucinations (Psychiatric disorders) | 1 (1)
Headache (Nervous system disorders) | 7 (7)
Hearing Impaired (Ear and labyrinth disorders) | 1 (1)
Hepatobiliary Disorders- Biliary Obstruction (Hepatobiliary disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 10 (12)
Hypertension (Vascular disorders) | 4 (16)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (4)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 2 (4)
Insomnia (Psychiatric disorders) | 3 (3)
Investigations (Left Axis Deviation) (Investigations) | 1 (1)
Lymphocyte Count Decreased (Investigations) | 1 (4)
Malaise (General disorders) | 1 (1)
Mucositis Oral (Gastrointestinal disorders) | 1 (1)
Muscle Cramp (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 5 (6)
Non-Cardiac Chest Pain (General disorders) | 1 (2)
Pain (General disorders) | 3 (3)
Paresthesia (Nervous system disorders) | 10 (16)
Peripheral Sensory Neuropathy (Nervous system disorders) | 2 (3)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Presyncope (Nervous system disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Psychiatric disorders - Vivid dreams (Psychiatric disorders) | 3 (3)
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 2 (3)
Rhinitis Infective (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Shingles (Infections and infestations) | 1 (1)
Sinus Bradycardia (Cardiac disorders) | 4 (8)
Sinus Tachycardia (Cardiac disorders) | 6 (14)
Skin and Subcutaneous Disorders (Blisters on Ear Lobes) (Skin and subcutaneous tissue disorders) | 1 (1)
Stomach Pain (Gastrointestinal disorders) | 3 (3)
Syncope (Nervous system disorders) | 2 (3)
Thromboembolic Event (Vascular disorders) | 3 (3)
Thrush (Infections and infestations) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Urinary Incontinence (Renal and urinary disorders) | 1 (1)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Weight Gain (Investigations) | 2 (2)
Weight Loss (Investigations) | 5 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-13): https://cdn.clinicaltrials.gov/large-docs/10/NCT04177810/Prot_SAP_000.pdf